CLINICAL TRIAL: NCT00179114
Title: Vanderbilt University Spasticity Management Program Evaluation Plan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Allergan (Industry); Medtronic (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMPEP-9.1
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-08-20 (Estimated); Status verified 2007-08

CONDITIONS: Spasticity
Keywords: Spasticity; Developmental Disabilities; Intrathecal baclofen (ITB); Botulinum Toxin Type A (Botox)
MeSH Terms: conditions — Muscle Spasticity; Developmental Disabilities | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum Toxin Type A
Drug: Intrathecal baclofen administered by the Medtronic SyncroMed(TM) pump (ITB)

SUMMARY:
People with severe developmental disabilities frequently have comorbidities that make providing care to them more difficult. Spasticity is one such comorbidity. It produces increased muscle tone that can cause stiffness in joints and bodily contortions that can interfere with all of the major types of care provided to participants. Typically, care areas include splinting, hygiene, dressing, transfers, positioning, ambulation, and engaging in other functional activities. Moreover, persons with spasticity often experience pain.

Typically, spasticity is managed by health care providers using a combination of the following therapies:

* Physical / occupational therapy (PT / OT)
* Oral medication
* Botox injections
* Intrathecal baclofen administered by the Medtronic SyncroMed pump (ITB)
* Orthopedic / neurological surgery

DETAILED DESCRIPTION:
As individuals are identified as appropriate participants for the Program and consent is obtained, the care team for each person, consisting of both medical and caregiver staff, will define up to three specific care area goals and related tasks for treatment. A comprehensive spasticity management program will then be developed for the individual. Clinical and outcome assessments at baseline and at follow-up will include measures of range of motion, global spasticity according to a modified Ashworth scale, and the time and number of staff required for the task. In addition, video will be obtained of caregivers performing each participant's care area tasks at baseline and follow-up to allow an independent external reviewer to judge task difficulty. Treatment will be provided as outlined by the spasticity management plan. Follow-up evaluations will be conducted when the participant is at least one year from their initial Botulinum injection, or are one year post-implant for ITB participants. When the participant is exited from the study, Survey Physician will be asked to rate the overall impact of the Program on each of the individual's care area tasks.

ELIGIBILITY:
Inclusion Criteria:

* Adult with spasticity residing at Clover Bottom Developmental Center in Nashville, Tennessee.
* Spasticity must interfere with daily functioning.
* Care team must be able to identify at least one treatment goal for the potential participant.

Exclusion Criteria:

* Family or guardian is unwilling to provide written informed consent.
* Spasticity does not interfere with patient's day-to-day care.
* Staff who provide daily care are unable to identify a clear treatment goal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-08; Study Completion 2006-02

PRIMARY OUTCOMES:
Total time (in seconds) spent by caregivers to complete a defined care area task at one year followup.
Categorical rating by blinded, independent reviewer of baseline and one-year care area task videos.

SECONDARY OUTCOMES:
Range of motion score for each care area goal, assigned by physical therapist and compared at baseline vs. one-year followup.
Differences in the number of hospital admissions 12 months pre- and 12 months post-program.
Differences in costs associated with caregiving 12 months pre- and 12 months post-treatment.
Difference in Physician's global assessment of spasticity at baseline and one-year followup.

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, MD, Principal Investigator — Vanderbilt University Department of Neurology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States